CLINICAL TRIAL: NCT07289984
Title: Correlation Between Diagnostic Nerve Block Response and Cryoneurolysis Outcome in Chronic Musculoskeletal Disorders and Spasticity
Acronym: CRYONIC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UniversitairZB25428; 25428 (Other: UniversitairZB)
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-11

CONDITIONS: Spasticity; Chronic Musculoskeletal Pain; Cryo Analgesia; Cryoablation
MeSH Terms: conditions — Muscle Spasticity | interventions — Cryosurgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chronic musculoskeletal pain group (Experimental)
  Interventions: Procedure: cryoablation

INTERVENTIONS:
Procedure: cryoablation — Cryoneurolysis

SUMMARY:
The clinical study is titled the CRYONIC PROTOCOL, which stands for Cryotherapy for Neurolysis In Chronic Pain and spasticity. It is structured as a prospective, multi-cohort observational study.

Purpose of the Study:

The overarching purpose of the CRYONIC PROTOCOL study is to assess the Correlation Between Diagnostic Nerve Block Response and Cryoneurolysis Outcome in Chronic Musculoskeletal Disorders and Spasticity. The study focuses on evaluating the effectiveness of ultrasound-guided peripheral nerve cryoneurolysis, a minimally invasive technique that uses extreme cold to induce temporary nerve blocks, for patients with treatment-resistant chronic musculoskeletal pain and spasticity.

The study also seeks to determine if cryoneurolysis itself leads to meaningful improvements in both pain intensity and functional ability in the included patient cohorts (those with chronic musculoskeletal pain or spasticity)

ELIGIBILITY:
Inclusion Criteria:

* Be over 18 year old
* Adults (> 18y) with either chronic musculoskeletal pain (> 3 months; average NRS > 5/10) or painful/functionally limiting spasticity
* Have a clinical stable condition, > 3months
* Any medications must be maintained on a stable schedule- Able to understand study instructions and provide informed consent (ICF) in French or Dutch.Provide written informed consent

Exclusion Criteria:

* Contraindication to cryoneurolysis such as a diagnosis of cryoglobulinemia, paroxysmal cold haemoglobinuria, cold urticaria, Raynaud's disease, any form of peripheral neuropathy, open and or infected wounds of the affected limb
* Patient's refusal to give consent to the procedure or to use of their data for research purposes.
* Ongoing local or systemic infection before the procedure.
* Predominantly neuropathic pain of the upper extremity as assessed with the Pain Detect questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2030-05-01 (Estimated); Study Completion 2031-08-01 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS) | 3 months
  Correlation between diagnostic nerve bloc and cryoneurolysis

SECONDARY OUTCOMES:
2-Minute Walk Test (2MWT) | 3 months
  A functional test measuring walking endurance (distance walked in 2 minutes); a practical measure of ambulatory capacity
Timed Up and Go | 3 months
  Measures the time taken to stand from a chair, walk 3m, turn, return, and sit, capturing basic mobility, balance, and fall risk
Passive Range of Motion | 3 months
  Joint angle measurement using a goniometer at the treated joint(s)
Goal Attainment Scaling | 3 months
  An individualized, patient-centered goal measure; goals are pre-defined and scored on a 5-point scale
Modified Tardieu Scale | 3 months
  Assesses spasticity across velocities; considered to have better construct validity for velocity-dependence than MAS
Modified Ashworth Scale | 3 months
  Clinician-rated 6-point ordinal scale quantifying muscle tone (resistance to passive movement)
Oswestry Disability Index (Low Back Pain) | 3 months
  Measures disability related to low back pain across 10 items focused on daily functioning
Shoulder Pain and Disability Index (Shoulder) | 3 months
  A self-administered questionnaire consisting of 13 items (5 for pain, 8 for disability) scored from 0 to 10
Disabilities of the Arm, Shoulder, and Hand (Arm/Shoulder) | 3 months
  A 30-item questionnaire evaluating upper limb function and symptoms
Hip Disability and Osteoarthritis Outcome Score (Hip) | 3 months
  Assesses hip-related pain, symptoms, activities of daily living, and QoL across five subscales (higher scores indicate better outcomes)
Knee Injury and Osteoarthritis Outcome Score (Knee) | 3 months
  Measures knee-related outcomes across five domains, including pain, symptoms, activities of daily living, and QoL
Work Ability Index | 3 months
  A 10-item questionnaire evaluating current work ability compared with the lifetime best, considering physical and mental demands and the impact of existing diseases
Medication Quantification Scale (Version III) | 3 months
  A validated tool to quantify the overall burden of pain medication based on pharmacological class, risk, and dose
Pain Self-Efficacy Questionnaire | 3 months
  Measures a patient's confidence in performing daily activities despite pain (10 items, scored 0 to 6)
Tampa Scale for Kinesiophobia (11 items) | 3 months
  Assesses fear of movement or (re)injury; higher scores (11 to 44) indicate more kinesiophobia
EuroQol 5 Dimensions, 5 Levels | 3 months
  A standardized instrument measuring general health status across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression
Patient-Reported Outcomes Measurement Information System - 29 items | 3 months
  Evaluates seven health domains, including physical function, anxiety, fatigue, and sleep disturbance
Brief Pain Inventory | 3 months
  Assesses both pain severity (scale 0-10) and the interference of pain with daily activities

IPD SHARING:
Plan to Share IPD: No